CLINICAL TRIAL: NCT06241222
Title: Origin of the Neonatal Gut Microbiota and Probiotic Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Zhe Li, Principal Investigator, Third Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: [2019]no.11EthicsCommittee
Record Dates: First submitted 2024-01-17; First posted 2024-02-05 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2024-07

CONDITIONS: Microbiota

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (No Intervention): pregnancies in control group need no intervention.
- probiotics group (Experimental): pregnancies in probiotics group need probiotics management
  Interventions: Drug: Probiotic Blend Oral Tablet

INTERVENTIONS:
Drug: Probiotic Blend Oral Tablet — In our study, fourteen pregnant women were randomly assigned to the probiotic group, and the rest were assigned to the control group. After enrollment, pregnant women in the probiotic group received a combination of living Bifidobacterium longum (5 ∗ 106 CFU), Lactobacillus delbrueckii bulgaricus (5 ∗ 105 CFU) and Streptococcus thermophilus (5 ∗ 105 CFU) tablets produced by Neimengu Shuangqi Pharmaceutical Co., Ltd. Pregnant individuals in the probiotic group were administered two tablets twice a day (2 g/d) until natural delivery
  Arms: probiotics group

SUMMARY:
This study aim to evaluate the composition and origin of the neonatal gut microbiota after birth and Probiotic intervention. Samples were obtained from a total of 30 pregnant individuals and their offspring, divided into control group and porbiotics group. Postpartum human milk and infant fecal specimens were collected for a period of 6 months. The samples were analyzed using 16S rRNA amplicon sequencing of the V3-V4 region to evaluate the microbial composition. The Shannon index, Simpson index and nonmetric multidimensional scaling were used to evaluate the diversity of the microbiota, while the co-occurrence network and LEfSe were used to evaluate the characteristics of the microbiota of pregnancies and their infants in each groups.

DETAILED DESCRIPTION:
Study design and participants A total of 30 samples were obtained from pregnant individuals receiving antenatal care at the 1st Affiliated Hospital of Jinan University. Informed consent was obtained from pregnant women (at least 32 gestational weeks) who met the inclusion criteria. Newborns were followed until 14 days after natural delivery. Pregnant inclusive criteria were: 1. Chinese woman who is pregnant with a single fetus; 2. First pregnancy and term delivery. Newborns' inclusive criteria were: 1. Normal weight (>2500 g, <4000 g); 2. Term Infant (>37 weeks, <42 weeks). 3. Natural birth. Pregnanct exclusive criteria were: 1. Gastrointestinal disease or family history; 2. Vaginitis before pregnancy; 3. Antibiotic usage during pregnancy; 4. Hypertension, Diabetes Mellitus, Hyperthyroidism, Hypothyroidism, Autoimmune Disease, or Other Endocrine and Metabolic Disease; 5. Gestational Hypertensive Disease, Gestational Diabetes Mellitus or Other Gestational Disease; 6. Transfusion History, Organ Transplantation History or Immunotherapy History. Newborn's exclusive criteria were: 1. Abnormal weight (>4000 g, <2500 g); 2. With Congenital Diseases;3. Intrapartum Fetal Complication.

Probiotic management In the investigators' study, fourteen pregnant women were randomly assigned to the probiotic group, and the rest were assigned to the control group. After enrollment, pregnant women in the probiotic group received a combination of living Bifidobacterium longum (5 ∗ 106 CFU), Lactobacillus delbrueckii bulgaricus (5 ∗ 105 CFU) and Streptococcus thermophilus (5 ∗ 105 CFU) tablets produced by Neimengu Shuangqi Pharmaceutical Co., Ltd. Pregnant individuals in the probiotic group were administered two tablets twice a day (2 g/d) until natural delivery, and those in the control group took no pills.

Fecal, vaginal secretion, placental, and meconium collection Fecal collection Feces from pregnant patients were collected twice-between weeks 32 and 34 and before natural labor. Feces collected at weeks 32-34 were collected internally, thereby avoiding contamination with foreign material. The feces were stored in a domestic refrigerator and transferred to the laboratory freezer at -80 ºC for 24 hours. Feces collected before labor were obtained in the hospital and transferred to the laboratory freezer within 30 min of collection.

Vaginal secretion collection Vaginal secretions were collected twice between weeks 32 and 34 and before natural labor. The pregnant woman was asked to not engage in sexual behavior, clean the vulva, clean the vagina, or use vaginal medicine within 48 hours before sample collection. Vaginal secretions before natural labor were collected before membrane rupture occurred. The samples were transferred to the laboratory freezer within 30 min of collection, thereby avoiding contamination by foreign material.

Placenta collection Placenta samples ranging from the entire umbilical cord to 3 cm were collected by stripping the amniotic membrane after natural birth. The blood was rinsed with sterile saline. Four to six pieces of placenta were sampled from the fetal surface. Each piece had a volume of approximately 1 cm3. The placenta sample was transferred to the laboratory freezer within 30 min of collection.

Meconium collection Meconium was collected three times on the 1st day, the 3rd day, and the 14th day after natural delivery On the 1st day and 3rd day, meconium was collected internally, thereby avoiding contamination with foreign material in the hospital, and was transferred to the laboratory freezer within 30 min of collection. On the 14th day, meconium was collected, stored in a domestic refrigerator, and then transferred to a laboratory freezer within 24 hours of collection.

When infants were 6 months old, postpartum milk was collected by two full-time members of the research group. The human milk samples were collected according to a standardized protocol. Before collecting the samples, the nursing mothers were required to clean the nipple and areola with soap and water. A total sample volume of 6 ml was collected in a sterile tube. Additionally, infant fecal samples were collected at the 6th month postpartum. After collection, the samples were stored with dry ice for transportation to the laboratory immediately. Upon arrival at the laboratory, the samples were briefly thawed to allow for accurate aliquoting. Each sample was then divided equally into smaller frozen storage tubes. The divided samples were promptly refrozen and stored in a freezer at -80°C within 4 hours after collection. This process ensured that the samples were handled with minimal temperature fluctuations to preserve their integrity.

Fecal samples from the infants were collected internally in sterile and dedicated collecting boxes, thereby avoiding any contamination with foreign material. These samples were stored in a domestic freezer (-20°C) and transferred to a laboratory freezer at -80°C within 24 hours using a cryogenic transport container to ensure they remained frozen during the transfer.

ELIGIBILITY:
Pregnant inclusive criteria were:

1. Chinese woman who is pregnant with a single fetus;
2. First pregnancy and term delivery.

Newborns' inclusive criteria were:

1. Normal weight (>2500 g, <4000 g);
2. Term Infant (>37 weeks, <42 weeks).
3. Natural birth.

Pregnancy exclusive criteria were:

1. Gastrointestinal disease or family history;
2. Vaginitis before pregnancy;
3. Antibiotic usage during pregnancy;
4. Hypertension, Diabetes Mellitus, Hyperthyroidism, Hypothyroidism, Autoimmune Disease, or Other Endocrine and Metabolic Disease;
5. Gestational Hypertensive Disease, Gestational Diabetes Mellitus or Other Gestational Disease;
6. Transfusion History, Organ Transplantation History or Immunotherapy History.

Newborn's exclusive criteria were:

1. Abnormal weight (>4000 g, <2500 g);
2. With Congenital Diseases;3. Intrapartum Fetal Complication.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
16S rRNA amplicon sequencing of the V4 region | 12 months
  Difference analysis of each group was performed. All the measurement data are presented as the mean ± standard error. Assessments of Operational Taxonomic Units differences in the probiotic group and control group were performed using independent sample t tests, and P < 0.05 was considered to indicate statistical significance. Other outcomes were analyzed using multiple linear regression. All data were analyzed using SPSS 23.0 statistical software (SPSS, Inc., Chicago, IL, USA).

CONTACTS AND LOCATIONS:
Locations (1):
- Zhe Li, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chen Y, Li Z, Tye KD, Luo H, Tang X, Liao Y, Wang D, Zhou J, Yang P, Li Y, Su Y, Xiao X. Probiotic Supplementation During Human Pregnancy Affects the Gut Microbiota and Immune Status. Front Cell Infect Microbiol. 2019 Jul 16;9:254. doi: 10.3389/fcimb.2019.00254. eCollection 2019. PMID 31380297
- [Background] Yang P, Li Z, Tye KD, Chen Y, Lu T, He Z, Zhou J, Xiao X. Effects of an orally supplemented probiotic on the autophagy protein LC3 and Beclin1 in placentas undergoing spontaneous delivery during normal pregnancy. BMC Pregnancy Childbirth. 2020 Apr 15;20(1):216. doi: 10.1186/s12884-020-02905-z. PMID 32295534
- [Background] Huang T, Li Z, Tye KD, Chan SN, Tang X, Luo H, Wang D, Zhou J, Duan X, Xiao X. Probiotic supplementation during pregnancy alters gut microbial networks of pregnant women and infants. Front Microbiol. 2022 Dec 1;13:1042846. doi: 10.3389/fmicb.2022.1042846. eCollection 2022. PMID 36532501
- [Derived] Meng L, Fan G, Xie H, Tye KD, Xia L, Luo H, Tang X, Huang T, Lin J, Ma G, Xiao X, Li Z. Maternal-to-neonatal microbial transmission and impact of prenatal probiotics on neonatal gut development. J Transl Med. 2025 Oct 30;23(1):1198. doi: 10.1186/s12967-025-07293-6. PMID 41168767
- [Derived] Ma G, Li Y, Tye KD, Huang T, Tang X, Luo H, Wang D, Zhou J, Li Z, Xiao X. The effect of oral probiotics in the last trimester on the human milk and infant gut microbiotas at six months postpartum: A randomized controlled trial. Heliyon. 2024 Aug 30;10(17):e37157. doi: 10.1016/j.heliyon.2024.e37157. eCollection 2024 Sep 15. PMID 39286230